CLINICAL TRIAL: NCT02491996
Title: The Efficacy of Cognitive-behavioral Therapy Focused on Desire-satisfaction for Treatment-seeking Disordered Gamblers
Brief Title: The Efficacy of Therapy Focused on Desire-satisfaction for Disordered Gamblers
Acronym: ETFDDG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kurihama Medical and Addiction Center (Other)
Responsible Party: Principal Investigator, Yasunobu Komoto, Chief of Treatment Unit for Gambling Disorder, Kurihama Medical and Addiction Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 223
Record Dates: First submitted 2015-02-27; First posted 2015-07-08 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Pathological Gambling
Keywords: desire model
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DTIG (Experimental): Outpatients who treated by DTIG at Outpatient Unit for Gambling Disorder of Kurihama Medical and Addiction Center
  Interventions: Behavioral: desire satisfaction-targeted intervention for disordered gamblers

INTERVENTIONS:
Behavioral: desire satisfaction-targeted intervention for disordered gamblers — This intervention consists of an initial psychiatric assessment, followed by psychoeducational approach based on desire satisfaction-targeted intervention by psychiatrists, and three group sessions based on CBT by psychologists. Patients with psychiatric comorbidities are treated with the appropriate pharmacological regimens.

SUMMARY:
The investigators proposed a desire satisfaction-targeted intervention for disordered gamblers (DTIG) due to the limitations of the abstinence-targeted intervention, which is based on the weak self-control relative to growing desire to gamble. This intervention model perceives loss of gambling control as a failure of strategy in which gambling is anticipated to fulfill various desires (i.e., desires for fame, money, and escapism). Therefore, the alternative behaviors to fulfill original desires directly become the main therapeutic purpose.

Materials and Methods: Outpatients who were primarily diagnosed as gambling disorder by the DSM-V were treated by DTIG. This method usually comprised 1 or 2 sessions, 60 minutes in duration, delivered by a psychiatrist. Participants were examined : 1) Basic background such as gender, age,; 2) medical variables such as the onset age, the duration of the problem gambling, psychiatric complications, motivation to quit gambling; 3) assessment of severity (DSM-5, SOGS and G-SAS); 4) Short prognosis; 6 months-outcome after intervention (problem gambling/ control gambling/ abstinence).

DETAILED DESCRIPTION:
Introduction

Gambling disorder is a public health problem characterized by persistent and recurrent maladaptive patterns of gambling. A prevalence rate was 0.4-2.0% worldwide. In Japan, gambling is common: the prevalence rate of disordered gamblers is estimated to be 5.5% of adults.Gambling disorder resulted in clinical and subclinical harms, which are depression, suicidal behaviors, legal involvement, occupational/ educational disruptions, financial and interpersonal difficulties.

Some psychological treatment studies indicate a benefit of active treatments compared to no treatment or wait-list control conditions. On the other hand, the accumulated evidence seems to suggest that interventions based on the CBT produce the most favorable outcomes.Nevertheless CBT is not yet recognized as a standard treatment for gambling disorder. What is the therapeutic insufficiency in CBT for gambling disorder? The fundamental aim of CBT, especially cognitive therapy for gambling disorder is to identify and correct irrational and unrealistic beliefs postulated to contribute to excessive gambling, which is usually the control over the outcome regardless of the randomness. However, although majority of disordered gamblers already understand that this belief is theoretically irrational, they cannot quit problem gambling. For recovery they may need not only cognitive changes in illusions of control but also motivated inner power such as desires.

Therefore the investigators assumed that disordered gamblers could not quit or control gambling because their original desires which had constructed pathological craving for gambling had not been satisfied. Namely most important erroneous beliefs for which the investigators should target in CBT are ones concerning not the nature of gambling itself but original desires. The investigators thought this hypothesis focused on original desire with reference to the studies of natural recovery process.

In this study, in order to reveal the efficiency of this intervention more clearly, for disordered gamblers the investigators compared a six months-outcome between this intervention, which we named a "desire satisfaction-targeted intervention for gambling disorder" (DTIG), and an ordinary abstinence-targeted intervention.

Methods:

Participants Subjects are outpatients who are treated by DTIG at Outpatient Unit for Gambling Disorder of Kurihama Medical and Addiction Center in Japan. This intervention consists of an initial psychiatric assessment, followed by psychoeducational approach based on desire satisfaction-targeted intervention by psychiatrists, and three group sessions based on CBT by psychologists. Patients with psychiatric comorbidities are treated with the appropriate pharmacological regimens.

All are over 20 years of age and meet Diagnostic and Statistical Manual of Mental Disorders 5thed. (DSM-5) criteria for a diagnosis of gambling disorder. 2) The investigators exclude patients with acute psychotic symptoms including manic symptoms or cognitive impairment that can compromise their ability to complete the research questionnaires.

This investigation is carried out in accordance with the Declaration of Helsinki, and going to be approved by the ethical committee of Kurihama Medical and Addiction Center. All subjects should be provided written informed consent.

Procedure

Participants are examined as follows at the first hospital visit:

1. Basic and medical background such as gender, age, married or not, educated beyond twelve years or not, employed or not, addiction-related family history (defined as a second-degree or closer family member with an addictive disorder), crime history, suicide history, current psychiatric complications;
2. Gambling-related variables such as the age of gambling onset, the age of problem-gambling onset, time lag between gambling onset and the onset of problematic gambling (time lag), the duration of the problem gambling, predominant gambling activity (non-strategic or not), total amount of debt, method of debt management (bankruptcy or not), Attendance at Self Help Group, motivation to quit gambling;
3. Assessment of severity such as the number of items in DSM-5, scores of South Oaks Gambling Screen (SOGS) 23) and the Gambling Symptom Assessment Scale (G-SAS) 15) ;
4. Outcome concerning gambling behavior in 3 and 6 months after DTIG.

Assessment of Severity Severity of gambling disorder is measured using the above three reliable and valid instruments.

1. DSM-5: The standard of severity is defined in the DSM-5 based on the number of items that are met: 4-5 is mild, 6-7 is moderate, and 8-9 is severe.
2. SOGS: 20-item self-report questionnaire providing a cut-off score for pathological gambling using DSM criteria. The accepted cut-off point for problem gambling is 5, with higher scores denoting more severe gambling problems.
3. G-SAS: 12-item self-report scale examining gambling urges, thoughts, and behaviors during the previous week.

Assessment of Outcome The investigators ask participants two questions concerning gambling behaviors 3 months and 6 months after intervention by mail or telephone, which are "Did participants gamble during this period (three or six months)?" and "Did some troubles with gambling happen during this three months if participants gambled?" The outcome is distinguished on a 3-stepped degree through the above two questionnaires; (keeping abstinence continuously / continuing gambling, but no problem during this three months / keeping problem gambling continuously). In this study, problem gambling was defined as "gambling accompanied by monetary, occupational/educational, familial and legal problem such as debts, absence, marital crisis and embezzlement etc."

Desire satisfaction-targeted intervention for gambling disorder (DTIG) The investigators have performed DTIG instead of ordinary abstinence-targeted intervention. In this intervention, whether patients currently gamble or not is once shelved. This intervention consists of three steps;

1. Identify original desires, which have been covered by intensive craving for gambling.
2. Aim to satisfy only a single desire if you hope to continue gambling.
3. Search and try alternative behaviors which directly satisfy the original desires.

One or two psycho-educational sessions based on above three steps were performed by psychiatrists (one session usually needs 30-60 minutes). A worksheet is utilized to progress this intervention smoothly.

Additionally three psycho-educational sessions are performed by psychologists to help to discover owns' desires (one session usually needs 60 minutes). These themes are "the total amounts of lost money", "advantage and disadvantage in gambling" and "alternative behaviors instead of gambling".

Statistical analysis Data entry and statistical analysis were performed using Microsoft ExcelⓇ 2010. A Pearson correlation analysis was used to assess correlations between outcome (abstinence / controlled gambling / problem gambling) and other variables in DTIG group. To identify the independent predictors of outcome, multiple stepwise backward linear regression analysis was used and an analysis of variance for the full regression models was performed.

These analyses were repeated using all participants (intention-to-treat analysis: ITT). Therefore cases that dropped out of the following system were set as cases that continued problem gambling (worst cases analysis). Statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were outpatients who are treated by DTIG at Outpatient Unit for Gambling Disorder of Kurihama Medical and Addiction Center in Japan. This intervention consists of an initial psychiatric assessment, followed by psychoeducational approach based on desire satisfaction-targeted intervention by psychiatrists, and three group sessions based on CBT by psychologists. Patients with psychiatric comorbidities are treated with the appropriate pharmacological regimens.

All were over 20 years of age and met Diagnostic and Statistical Manual of Mental Disorders 5thed. (DSM-5) criteria for a diagnosis of gambling disorder.

Exclusion Criteria:

* We exclude patients with acute psychotic symptoms including manic symptoms or cognitive impairment that could compromise their ability to complete the research questionnaires.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Severity of gambling | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Naruse Mental Clinic, Machida, Tokyo, Japan